CLINICAL TRIAL: NCT01442935
Title: Phase II Multicentric Randomized Trial, Evaluating the Best Protocol of Chemotherapy, Associated With Targeted Therapy According to the Tumor KRAS Status, in Metastatic Colorectal Cancer (CCRM) Patients With Initially Non-resectable Hepatic Metastases
Brief Title: Chemotherapies Associated With Targeted Therapies on the Resection Rate of Hepatic Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 14 / ACCORD 21/0905; 2009-012813-22 (EudraCT Number)
Record Dates: First submitted 2011-08-10; First posted 2011-09-29 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: Adenocarcinoma; Non-resectable hepatic metastases; First-line treatment
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A1 : Folfiri + targeted therapy (Active Comparator): Every 2 weeks :
  * irinotecan 180 mg/m² D1
  * Folinic acid 400 mg/m² D1
  * 5FU 400 mg/m² bolus
  * 5FU 2400 mg/m² infusion over 46 h, D1
  And targeted therapy in function of Kras:
  * For mutated Kras = bevacizumab: 5 mg/kg IV on D1 of each cycle of chemotherapy, every 14 days
  * For non-mutated Kras = cetuximab : 500 mg/m² IV, on D1 of each cycle of chemotherapy, every 14 days.
  Interventions: Drug: Folinic Acid; Drug: 5-FU; Drug: Irinotecan; Drug: Bevacizumab; Drug: Cetuximab
- Arm A2 : Folfox 4 + targeted therapy (Active Comparator): Every 2 weeks :
  * oxaliplatin 85 mg/m² D1
  * Folinic acid 400 mg/m² D1
  * 5FU 400 mg/m² bolus
  * 5FU 2400 mg/m² infusion over 46 h, D1
  And targeted therapy in function of Kras:
  * For mutated Kras = bevacizumab: 5 mg/kg IV on D1 of each cycle of chemotherapy, every 14 days
  * For non-mutated Kras = cetuximab : 500 mg/m² IV, on D1 of each cycle of chemotherapy, every 14 days.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-FU; Drug: Bevacizumab; Drug: Cetuximab
- Arm B : Folfirinox + targeted therapy (Experimental): Every 2 weeks :
  * oxaliplatin 85 mg/m² D1
  * irinotecan 150 mg/m² D1
  * Folinic acid 400 mg/m² D1
  * 5FU 400 mg/m² bolus
  * 5FU 2400 mg/m² infusion over 46 h, D1. From D7 to D12, prophylactic G-CSF such as Granocyte® will be administered.
  And targeted therapy in function of Kras:
  * For mutated Kras = bevacizumab: 5 mg/kg IV on D1 of each cycle of chemotherapy, every 14 days
  * For non-mutated Kras = cetuximab : 500 mg/m² IV, on D1 of each cycle of chemotherapy, every 14 days.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-FU; Drug: Irinotecan; Drug: Bevacizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Oxaliplatin — 85mg/m² over 120 mn every 2 weeks up to progression or toxicity
  Arms: Arm A2 : Folfox 4 + targeted therapy; Arm B : Folfirinox + targeted therapy
Drug: Folinic Acid — 400mg/m² over 120 mn every 2 weeks up to progression or toxicity
Drug: 5-FU — 400mg/m² in bolus, then 2400mg/m² over 46 h every 2 weeks up to progression or toxicity
  Other Names: 5-Fluoro uracil
Drug: Irinotecan — 180mg/m² over 90 mn every 2 weeks up to progression or toxicity
  Arms: Arm A1 : Folfiri + targeted therapy
Drug: Irinotecan — 150mg/m² over 30-90 mn every 2 weeks up to progression or toxicity
  Arms: Arm B : Folfirinox + targeted therapy
Drug: Bevacizumab — 5mg/kg over 90 mn every 2 weeks up to progression or toxicity
Drug: Cetuximab — 500mg/m² over 90 mn every 2 weeks up to progression or toxicity

SUMMARY:
The main objective is to compare resection rates (R0 or R1) for hepatic metastases in the experimental arm (tri chemotherapy plus targeted therapy) versus the control arm (bi chemotherapy plus targeted therapy); in both arms the targeted therapy is selected according to K-Ras status of the patient's tumor.

The secondary objectives are to evaluate the objective response rate (CR and PR) after 4 cycles of treatment, according the RECIST V1.1 evaluation scale.

* the rate of complete remission (CR) at 6 months after the last study treatment (hepatic surgery or last chemotherapy cycle).
* the specific rates of resection R0, R1, R2.
* the complete pathological response Rate,
* the relapse-free survival rate in (R0 or R1) resected patients,
* the response duration in non-resected patients,
* the toxicity according to CTC AE V4 scale except for the neurotoxicity that will be evaluated with the Levi scale,
* the post operative complications using the DINDO classification,
* the progression-free survival (PFS) and overall survival (OS).

The objectives of the biological study are:

* to evaluate tumor-related predictive factors such as somatic mutations (KRAS, BRAF, TP53) and genetic amplification related factors (EGFR),
* to evaluate patient-related predictive factors in connection with genetic polymorphisms (Fc gamma and VEGF receptors),
* to evaluate ADCC activity via immunohistochemistry in order to analyze the lympho free and progression-free survival,
* to study circulating of tumor cells as prognostic factor for metastatic colorectal cancer, non- resectable at presentation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma,
* Primary tumor of the colon or rectum, resectable or resected at least 3 weeks before randomization or 4 weeks before the beginning of the study treatment,
* Metastatic disease with synchronous or metachronous (> 3 months after diagnosis of the primary tumor) hepatic metastasis,
* Non-resectable (with respect to curative intent) hepatic metastasis at presentation. This criterion must be validated by both a surgeon and a radiologist during the RCP (Multidisciplinary cancer case presentation committee) patient's evaluation meeting (either technically non-resectable metastases (absolute contraindication): i.e. impossibility to resect all metastases in a single operation while preserving at least 30% of healthy liver tissues and/or impossibility to preserve the portal vein and hepatic artery homolateral to the liver or a portal pedicle, or due to oncological non-resectability (relative contraindication): presence of > 5 nodules and bilateral invasion),
* Hepatic metastases, without spread to other sites except in case of ≤ 3 resectable pulmonary metastases of diameter < 2 cm, detected by thoracic scanner,
* K-Ras status determined before randomization,
* Measurable disease according to the RECIST V1.1 criteria,
* No prior treatment of the hepatic metastases,
* Previous 5FU +/- oxaliplatin-based adjuvant chemotherapy administered after colorectal tumor resection is authorized if complete more than 1 year before,
* Age ≥ 18 & ≤ 75 years
* Performance status : ECOG 0 or 1,
* Life expectancy ≥ 3 months,
* Hemoglobin ≥ 9 g/dl,
* Polynuclear neutrophiles ≥ 1500/mm3,
* Platelets ≥ 100 000 mm3,
* Creatinemia ≤ 135 µmol/l (1,35 mg/dl)
* Total bilirubin ≤ 1.25 times the Upper Limit of Normal (ULN).
* Hepatic enzymes ASAT and ALAT < 5 x ULN,
* Negative pregnancy test for women of child-bearing age,
* Information given to the patient and signed informed consent,
* Public Health insurance coverage.

Exclusion Criteria:

* Non metastatic and/or non measurable disease according to the RECIST v1.1 criteria.
* Non-resectable primary tumor (e.g.: T4 tumors) or incomplete resection R2.
* History of intestinal inflammatory disease.
* Specific contraindication to any of the study treatments.
* Patient who have previously received anti-EGFr (e.g., cetuximab) or anti-VEGF monoclonal antibody treatment (e.g., bevacizumab) or treatment with irinotecan.
* History of cancer considered as not cured.
* Stroke/CVA or pulmonary embolism within 6 months before inclusion.
* Significant concomitant disease such as: coagulopathy, respiratory or cardiac congestive insufficiency, non-medically controlled/unstable angina pectoris, myocardial infarction within 6 months prior to study entry, arterial hypertension and uncontrolled arrhythmia, severe infections.
* Clinical neuropathy, grade ≥1.
* Patient already included in another therapeutic trial using an experimental molecule.
* Pregnant women or women who might become pregnant during the study or lactating women.
* Men or women who can procreate and who do not abide with the use of a contraceptive means.
* Persons kept in detention or incapable of giving consent
* Patient unwilling or unable to comply with the medical follow-up required by the trial because of geographic social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
The main objective is to compare resection rates (R0 or R1) for hepatic metastases | at least 4-6 weeks after the end of chemotherapy
  Number of patients (%) with hepatic metastases R0 or R1 resection.

SECONDARY OUTCOMES:
The objective response rate (CR and PR) after 4 cycles of treatment | after 8 weeks
  The objective response rate (CR and PR) will be evaluated by the investigator with RECIST v1.1 criteria after 4 cycles. Patients with symptoms suggestive of disease progression will have a tumoral evaluation when symptoms will occur
Complete remission rate (CR) 6 months after the last study treatment (hepatic surgery or last chemotherapy cycle) | 6 months
  Number of patients (%) with complete remission (CR) at 6 months after the last study treatment (hepatic surgery or last chemotherapy cycle)
Specific resection rates R0/R1/R2 | 24 weeks
  Specific resection rates (%) R0/R1/R2 is the rate of patients with a R0, R1 or R2 resection.
Complete pathological response | 24 weeks
  Number of patients with Complete pathological response, defined as the absence of tumoral residues after the last chemotherapy cycle. It will be evaluated on liver resection piece, based on total or complete tumor necrosis in all tumor nodules
Toxicity of treatment | Every 2 weeks
  Tolerance of the treatment will be based on toxicities of evaluated products by clinical and biological measurements (NCIC/CTC (CTCAE V4) criteria, except for peripheral neuropathy toxicity (Lévi scale)
Post operatory complications | after 4 weeks
  Each post operatory complications (Hemorrhage, fistula, insufficiency, heart failure,..) will be graduated using Dindo classification (2004)
Progression-free survival (PFS) | 8 months
  Progression-free survival is defined as the time from randomization to progression (RECIST v1.1 criteria) or death. Patients alive without progression will be censored at the last follow-up.
Overall survival (OS) | 14 months
  Overall survival is defined as the time from randomization to death any cause or last follow-up news for patients alive (censored data).

CONTACTS AND LOCATIONS:
Overall Officials: Marc YCHOU, Pr, Principal Investigator — Centre Val d'Aurelle; Eric FRANCOIS, Dr, Principal Investigator — Centre Antoine Lacassagne, Nice; Laurent MINEUR, Dr, Principal Investigator — Institut Ste Catherine-AVIGNON; Olivier BOUCHE, Pr, Principal Investigator — CHU de Reims; Driffa MOUSSATA, Dr, Principal Investigator — Centre hospitalier Lyon Sud-PIERRE BENITE; Rosine GUIMBAUD, Pr, Principal Investigator — Centre hospitalier Rangueil-TOULOUSE; Roger FAROUX, Dr, Principal Investigator — CHD Vendée -LA ROCHE SUR YON; Karine BOUHIER-LEPORRIER, Dr, Principal Investigator — CHU Côte de Nacre-CAEN; Alice GAGNAIRE, Dr, Principal Investigator — CHU Dijon - Hôp. Du Bocage; Yves BECOUARN, Dr, Principal Investigator — Institut Bergonié Bordeaux; François GHIRINGHELLI, Dr, Principal Investigator — Centre G. F. Leclerc-DIJON; Rosine GUIMBAUD, Pr, Principal Investigator — Centre hospitalier Purpan-TOULOUSE; Gaël DEPLANQUE, Dr, Principal Investigator — Centre Hospitalier Saint-Joseph-PARIS; Julien FORESTIER, Dr, Principal Investigator — Hôpital Edouard Herriot-LYON; Pascale MARIANI, Dr, Principal Investigator — Institut Curie Paris; Jean-Louis LEGOUX, Dr, Principal Investigator — CHR d'Orléans - La Source; Cédric LECAILLE, Dr, Principal Investigator — Polyclinique de Bordeaux Nord; Marie-Pierre GALAIS, Dr, Principal Investigator — Centre François Baclesse-CAEN; Philippe HOUYAU, Dr, Principal Investigator — Clinique Claude Bernard, Albi
Locations (1):
- Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Derived] Bidard FC, Kiavue N, Ychou M, Cabel L, Stern MH, Madic J, Saliou A, Rampanou A, Decraene C, Bouche O, Rivoire M, Ghiringhelli F, Francois E, Guimbaud R, Mineur L, Khemissa-Akouz F, Mazard T, Moussata D, Proudhon C, Pierga JY, Stanbury T, Thezenas S, Mariani P. Circulating Tumor Cells and Circulating Tumor DNA Detection in Potentially Resectable Metastatic Colorectal Cancer: A Prospective Ancillary Study to the Unicancer Prodige-14 Trial. Cells. 2019 May 28;8(6):516. doi: 10.3390/cells8060516. PMID 31142037